CLINICAL TRIAL: NCT00946140
Title: Motion Correction in Dynamic Contrast Enhanced MRI in Ovarian Cancer: A Pilot Study
Brief Title: Motion Correction in Dynamic Contrast Enhanced Magnetic Resonance Imaging (MRI) in Ovarian Cancer: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-132
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Ovarian Cancer
Keywords: Ovary; MRI; 08-132
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with ovarian cancer currently undergoing treatment: All of the patients will be treated per their treatment protocols by their physicians and they will be referred to this study for the DCE-MRI scans at baseline, within 24-48 hours of the start of the therapy, and within 6-8 weeks of the start of the therapy.
  Interventions: Procedure: DCE-MRI scans

INTERVENTIONS:
Procedure: DCE-MRI scans — Initially you will be given safety information about MRI scans and a questionnaire to determine your compatibility with the MRI scanner. For each patient, DCE-MRI data sets will be acquired three times - at baseline just prior to the start of the drug therapy, within 24-48 hours of the start of the therapy, and within 6-8 weeks of the start of the therapy.

SUMMARY:
The purpose of this study is to develop new image analysis method using Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE-MRI) for ovarian cancer. MRI is not currently part of the standard care for ovarian cancer. In this method, a contrast agent is used to make ovarian cancer visible during imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable disease with evidence of at least one uni-dimensionally measurable tumor (> 1 cm) by CT or MRI scan according to RECIST (Response Evaluation Criteria in Solid Tumors) that the tumor has not been initially treated with surgery or radiation therapy.
* Patients who will start treatment with bevacizumab combined with or without cytotoxic chemotherapy within 14 days from signing consent. Patients treated on an approved IRB therapeutic protocol for recurrent ovarian cancer with bevacizumab are eligible.
* Patients with histologically confirmed ovarian epithelial cancer including primary peritoneal and fallopian tube adenocarcinoma.
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception.
* Patients who are older than 21 years of age.
* Patients who are able to understand and sign informed consent.

Exclusion Criteria:

* Patients treated on an approved IRB therapeutic protocol with a blinded arm of bevacizumab or placebo are not eligible (IRB 07-078 and IRB 05-138).
* Patients with cardiac pacemakers.
* Patients with certain prosthetic devices and implants who are not compatible with the high magnetic field present in the DCE-MRI scanners.
* Patients who have experienced a prior adverse reaction to the gadolinium complex contrast agent used in DCE-MRI imaging and who don't meet criteria for creatinine and nephrogenic systemic sclerosis risk per guidelines of department of radiology.
* Patients prone to claustrophobia.
* Patients on dialysis.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the existing patient population at Gynecologic Medical Oncology Service at MSKCC. The patients meeting the eligibility criteria will be referred to DCE-MRI study by a physician in the GMO service at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Development of automated motion correction algorithms and new functional methods that permit use of DCE-MRI in primary or metastatic tumors of the ovaries. | 2 years

SECONDARY OUTCOMES:
Testing of new methods using the DCE-MRI data sets for comparing changes in tumor perfusion with and without motion correction post anti-angiogenic therapy in ovarian cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Gultekin, Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org